CLINICAL TRIAL: NCT03513146
Title: Impact of Oropharyngeal Administration of Mother's Milk Prior to Gavage Feeding on Hospital Acquired Neonatal Infection
Brief Title: Oropharyngeal Administration of Mother's Milk in Preterm Infants and Neonatal Infection
Acronym: OPAMM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University Children Hospital (Other)
Responsible Party: Principal Investigator, Nehad Nasef, Professor of Pediatrics, Mansoura University Children Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MS-15.09.03
Record Dates: First submitted 2018-04-19; First posted 2018-05-01 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Preterm Infant; Neonatal SEPSIS; Neonatal Feeding Disorder
MeSH Terms: conditions — Premature Birth; Neonatal Sepsis

STUDY DESIGN:
Intervention Model Description: Oropharyngeal Administration of mother's milk (OPAMM)
Who Masked: Outcomes Assessor
Masking Description: Microbiological assessment of bacterial colonization of the oropharyngeal cavity and the GIT will be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OPAMM group (Experimental): During the pre-feeding period, infants will receive mother's colostrum (to the maximum of 0.2 ml) by dropper to the oro-pharyngeal pouch, tongue and cheeks every 2 to 4 hours.
  When an infant fits the criteria to start enteral feeding, 0.2 ml of own mother's milk will be given by dropper to the oro-pharyngeal pouch, tongue and cheeks and the remaining amount will be given by the regular gavage feeding on intervals and amount regulated by the feeding protocol.
  This practice will be continued till the infants reach full oral feeding.
  Interventions: Procedure: Oropharyngeal Administration of Mother's Milk (OPAMM)
- Control Group (No Intervention): During the pre-feeding period, preterm infants will remain NPO. When an infant fits the criteria to start enteral feeding, own mother's colostrum or milk will be given by the regular gavage feeding on intervals regulated by the feeding protocol.
  This practice will be continued till the infants reach full oral feeding.

INTERVENTIONS:
Procedure: Oropharyngeal Administration of Mother's Milk (OPAMM) — 0.2 ml of own mother's milk will be given by dropper to the oro-pharyngeal pouch, tongue and cheeks and the remaining amount will be given by the regular gavage feeding on intervals and amount regulated by the feeding protocol
  Arms: OPAMM group

SUMMARY:
The protective effect of mother's milk and colostrum on oropharyngeal cavity is not achievable with gavage feeding. This may be increase the risk of colonization of the oropharyngeal cavity with pathogenic bacteria and subsequent increase in the risk of neonatal sepsis. We aim to study the impact of Oropharyngeal Administration of Mother's Milk (OPAMM) before gavage feeding on clinical outcome, bacterial colonization of the GIT of preterm infants with pathogenic bacteria. We also aim to study the immune-protective effect of OPAMM on the incidence of nosocomial sepsis.

DETAILED DESCRIPTION:
Preterm, very low Birth Weight (VLBW), infants are at increased risk of feeding intolerance as they have shorter GIT with lower digestive, absorptive and motility capabilities than those of full term infants. Intolerance to enteral feeding has been associated with abdominal distention, initiation of an inflammatory cascade, edema of the bowel, and subsequent development of necrotizing enterocolitis (NEC).

Oral feeding is the best and physiologic method for enteral nutrition of preterm infants. However, because of immaturity of suckling reflex and poor coordination between suckling and swallowing, gavage (oro-gastric or nasogastric tube feeding) has been used as an alternative method of enteral nutrition in preterm infants.

The gut of preterm infants is frequently colonized with pathogenic bacteria due to prematurity, increase gut mucosal permeability, delayed initiation of feeding, formula feeding, and frequent use of antibiotics. This pathogenic bacteria increase the chance of development of nosocomial acquired sepsis and NEC.

Mother's milk, particularly colostrum, is rich in cytokines and other immune agents that provide bacteriostatic, bacteriocidal, antiviral, anti-inflammatory and immunomodulatory protective agents against infection. Thus early gut priming and initiation of enteral feeding of preterm infants with mother's colostrum and milk decrease pathogenic bacterial colonization and subsequent development of sepsis and NEC.

During breast feeding, mother's milk comes in contact with the mouth and oro-pharyngeal pouch which, theoretically, stimulate both oropharyngeal receptors that improves the motility, secretory and absorptive ability of the GIT. Furthermore, anti-inflammatory and pro inflammatory cytokines, which are present abundantly in mother's colostrum and milk, may exert an immuno-protective effect when they come in contact with oropharyngeal as well as GIT mucosa.

We aim to study the impact of Oropharyngeal Administration of Mother's Milk (OPAMM) before gavage feeding on clinical outcome, bacterial colonization of the GIT of preterm infants with pathogenic bacteria. We also aim to study the immune-protective effect of OPAMM on the incidence of nosocomial sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants delivered at less than 32 weeks gestation and less than 1500 grams birth weight will be included in the study

Exclusion Criteria:

1. Preterm infants < 32 weeks gestation unable to be fed on own mothers' colostrum or milk.
2. Preterm infants with major congenital anomalies or chromosomal abnormalities.
3. Preterm infants delivered to mothers with confirmed chorioamnionitis
4. Preterm infants with confirmed early onset sepsis.

Ages: 1 Day to 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Hospital Acquired late onset neonatal sepsis | Neonatal care unit admission
  Culture proven neonatal sepsis acquired during neonatal care admission

SECONDARY OUTCOMES:
Colonization of the oro-pharyngeal pouch with pathogenic micro-organism | Neonatal care unit admission
  Throat swab will be taken at the start of the study and at the end of full enteral feeding.
Colonization of the GIT with pathogenic micro-organism | Neonatal care unit admission
  Stool culture will be taken at the start of the study and at the end of full enteral feeding.
Necrotizing enterocolitis | Neonatal care unit admission
  Bell's stage II of necrotizing enterocolitis
Ventilator associated pneumonia | Neonatal care unit admission
  Clinical and radiological evidence of Ventilator associated pneumonia

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Children Hospital, Al Mansurah, El Dakahlya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Panchal H, Athalye-Jape G, Patole S. Oropharyngeal Colostrum for Preterm Infants: A Systematic Review and Meta-Analysis. Adv Nutr. 2019 Nov 1;10(6):1152-1162. doi: 10.1093/advances/nmz033. PMID 31147686